CLINICAL TRIAL: NCT07175792
Title: Assessment of Perceptive Accuracy for Motor Performance in Persons With Multiple Sclerosis
Brief Title: Accuracy of Motor Performance Perception in Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Peter Feys, Prof. dr., Hasselt University
Other Study IDs: B1152024000009
Record Dates: First submitted 2025-08-19; First posted 2025-09-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Motor Performance; Task-specific; Perception; Multiple Sclerosis; Walking; Sit-to-stand; Inteoception
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with Multiple Sclerosis: Inclusion criteria: Age between 18 and 70 years old; a diagnosis of MS (2017 revisions of the McDonalds criteria); ability to walk for 6 minutes without rest and without the need of a walking aid; ability to repeatedly perform the sit to stand transitions on a standard chair (43cm seat height) without hand support. Additionally, no relapses >1 month preceding the start of the study.
  Exclusion criteria: cognitive impairment hindering understanding of study instructions, pregnancy, and musculoskeletal disorders in the lower limbs (not related to MS), cardiovascular red flags for exercise (screened with Physical Activity Readines Questionnaire), other diagnosis for neurological or metabolic disease limiting the full execution of the tests (eg. peripheral neuropathy altering the foot plantar sensibility).
- Healthy Controls: Age and sex matching is ensured within a five-year range per Healthy Contol.
  Exclusion criteria: cognitive impairment hindering understanding of study instructions, pregnancy, and musculoskeletal disorders in the lower limbs, cardiovascular red flags for exercise (screened with Physical Activity Readines Questionnaire), other diagnosis for neurological or metabolic disease limiting the full execution of the tests (eg. peripheral neuropathy altering the foot plantar sensibility).

SUMMARY:
The aim of this study is to characterize perceptive abilities in PwMS compared to controls when performing prolonged functional tasks such as walking and repeated standing from a seated position.

This study proposes primary and secondary research questions which will be tested in the context of two different newly designed experimental tasks and will be performed in maximum three days.

The self-reported beliefs over perceptive abilities and the performance in the experimental perceptive tasks will be compared between persons with multiple sclerosis and an equally sized group of age and gender matched healthy controls. The results of this study may uncover specific deficits in the MS population and will help in defining subgroups of patients with weaker perceptive capacities to gauge their motor performance and therefore in need for tailored interventions additional to the standard practice.

DETAILED DESCRIPTION:
For all work packages, the following information will be recorded from all participants in the first day: demographic data and PROMs of physical activity level [Godin Leisure-Time Exercise questionnaire], sleep quality [Pittsburgh Sleep Quality Index], self-efficacy [General and MS-specific Self-Efficacy scales], affectivity [Positive and Negative Affect Schedule], anxiety and depression [Hospital Anxiety and Depression Scale], habitual symptoms and fatigue [Checklist for Symptoms in Daily life, Brief Pain Inventory, Fatigue Scale for Motor and Cognitive Functions and Modified Fatigue Impact Scale], body and mobility perception [Multidimensional Assessment of Interoceptive Awareness (MAIA-2), Interoceptive Sensitivity and Attention Questionnaire (ISAQ), Postural Awareness Scale (PAS), Multiple Sclerosis Walking Scales, Falls Efficacy Scale] are recorded via secured digital surveys (CASTOR© Electronic Data Capture system). Symbol Digit Modalities Test (SDMT) for processing speed; Brief Visuospatial Memory Test (BVMT) for memory skills; Dual Joint Position Test (DJPT) for proprioception Timed 25-Foot Walk test (T25FW) for maximal walking speed; Test for the Sensory Interaction of Balance (for postural control; 6-Minutes Walking Test (6MWT, walking as far but safe during 6') and 30 seconds Chair Stand Test (30CST, completing as many STSs in 30 seconds) for specific walking and STS performance. IMUs are applied (APDM©, see below) and subjective state fatigue is measured before and after motor performance tasks using a Visual Analogue Scale (VAS, scoring from 0 to 10).

Work package 1a -Protocol: Participants will be familiarized with task-specific perceptual reporting methods. Standardized instructions are formulated in a neutral way to not bias participants' attention toward their symptoms. They will be instructed to report the time-points of perceived changes ("as soon as you perceive it"), either positive or negative, in quantitative or qualitative aspects of their motor performance: the speed or the smoothness of their self-motion. It is explained to the participants as 'a movement that happens in a continual fashion, without any interruptions'. To collect reports we designed a light portable haptic device fitting in the hand (shaped in a similar fashion as the Jamar hand-dynamometer®) and connected via Bluetooth® to a peak-detection Matlab© algorithm. Reports were given by a squeeze. To remove the signal noise produced by involuntary hand-grip forces, the threshold sensitivity of the sensor (i.e., minimum to save a report) will be set at 25% of the maximal hand-grip strength of the participant.

The first task involves a 6MWT at maximal walking speed in silence (eg. no information on time-on-test or verbal encouragements), while instructed to perceive fluctuations in either speed either smoothness (2 walking sessions, counterbalanced order) fluctuations and, as soon as they perceive a performance change, squeeze the sensor in the handheld device. The second task consists on repeated STS transitions: participants perform STSs at a fixed pace (one every ten seconds for six minutes), each one attempting to maximize speed, from a chair with normalized seat-height (lower leg length). Participants will use the handheld force sensor to indicate when variations are perceived during the task, comparing speed/smoothness (2 STS sessions, counterbalanced order) of consecutive STS transitions. Motor performance in the 2 tasks will be recorded with wearable sensors: 6 APDM© inertial motion units (2 over the dorsal part of the feet, 2 on the lower legs, 1 anterior to the sternum and 1 posterior to the fourth lumbar vertebra). The recordings allow for an objective comparison between reported and actual performance variations. Fatigue perception will be assessed before and after each session using the VAS. A brief interview will follow, asking participants to rate their confidence for having been accurate in detecting performance variations (on a scale from to 100) and to describe their own strategy: the sensory cues they relied on, for their reports.

-Work package 1b. "Imposed motor performance" WP1b assesses perceptive awareness for externally-imposed motor performance variations. After assessing perceptive sensitivity for performance variations in self-paced scenarios, we now focus on the quantification of subjects' perceptive accuracy using a real-time verbal reporting approach. Like in WP1a, we will use 2 tasks, walking and STS, with order counterbalanced at group level.

Protocol Walking task - Treadmill Participants will familiarize during a 10-minute supervised treadmill session with the moving belt, safety bars, and general usability. To determine a personalized speed range, participants will start walking at 50% of their maximal walking speed, calculated in their 6MWT overground performance as the highest 15-second moving average. They need to confirm if that is their comfortable treadmill walking speed. If not, adjustments will be made. Participants will see a vertical visual scale in front of them to indicate perceived variations: verbal descriptors will indicate walking speed, with 0% representing comfort and +100% representing maximal walking speed. Afterwards, they will be instructed to adapt their gait to continuous belt acceleration toward their maximal walking speed. This is as familiarization with their personalized range of speed: they will be informed about every 10th step on the VAS (0-100), experiencing how it feels to walk at those speed levels.

Participants will walk on a treadmill with the speed systematically increasing and decreasing within the predefined individual range. The task lasts 6 minutes, starting with 1 minute at the self-selected comfortable speed. Then, speed increases for all participants by 1.5 km/h in 15 steps (0.1 km/h each) over 150 seconds, never exceeding the participant's max walking speed. After a brief plateau, imposed speed is decreasing in the same manner over 150 seconds. Speed changes occur at randomly timed intervals of 5-15 seconds each while verbal reports are prompted and recorded every 10 seconds. The choice of a fixed range of imposed speed, with identical magnitude and timing of speed increments, was defined after piloting the experiment with PwMS and HC to ensure a standardized comparison of absolute speed changes between groups. In order to not alter the participants' gait pattern on the treadmill, we avoided the use of a safety harness, what was also not needed for PwMS with mild impairment. Also, to remove external cues as treadmill sound, we ask participants to wear noise cancelling headphones playing white noise.

Protocol STS task - Chair for Interoceptive Assessment n.0 (CIA0) To impose STS difficulty variations, we mounted a standard chair on a hydraulic system that allows real-time seat height adjustments while an infrared optical sensor continuously measures the distance from the ground, ensuring precise control. This setup enables dynamic and personalized STS assessments and training and we believe it may open new possibilities for rehabilitation and tele-rehabilitation. The baseline seat height will be individually normalized to each participant's lower leg length (measured as the distance from the ground to the inferior margin of the patella). To define a personalized range of imposed difficulty, the seat height will be adjusted between ±20% of this baseline, with the lowest height representing the most challenging condition. Participants will familiarize themselves with each STS level by performing transitions at different seat heights while being informed of their corresponding position on a vertical visual scale (every 10th step, ranging from 0% comfort to -100% minimal seat height).

Participants will perform STS transitions at a fixed pace and completing one repetition every 10 seconds, but always starting from a standing position, sitting down and immediately after shifting their weight on the chair stand up as quickly as possible. No specific instructions are given about the stand-to-sit phase, considered as part of the perceptive strategy. To ensure they rely solely on movement perception, they look straight ahead not receiving any feedback on seat height changes. During the stance phase in between STS repetitions, the seat height will be modified starting from the baseline (comfortable seat-height= lower leg length + its 20%) with fixed decrements (5% of lower leg length) but with randomized number of repetitions (0, 1 or 2) in between variations in seat height. The seat-height lowering will continue down to the personalized lowest seat-height (not having safety constraints in this case), stabilizing on that value before increasing toward the baseline height. After each repetition, participants will verbally report the number corresponding to their perceived difficulty level based on the pre-established scale.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years old
* ability to walk for 6 minutes without rest and without the need of a walking aid
* ability to repeatedly perform the sit to stand transitions on a standard chair (43cm seat height) without hand support

For People with Multiple Sclerosis group

* a diagnosis of MS (2017 revisions of the McDonalds criteria)
* no disease relapses >1 month preceding the start of the study

Exclusion Criteria:

* cognitive impairment hindering understanding of study instructions
* ongoing or suspected pregnancy
* musculoskeletal disorders in the lower limbs
* cardiovascular red flags for exercise (screened with Physical Activity Readines Questionnaire)
* other diagnosis for neurological or metabolic disease limiting the full execution of the tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 44 PwMS and 44 healthy controls will be recruited from the Flemish MS rehabilitation centers in Melsbroek (NMSC) and Pelt (Noorderhart RMSC), and as well from the REVAL research center in UHasselt. No economical compensation will be provided. We will search age and sex-matching healthy controls, considering a 5-year range per subject. After giving informed consent, demographics of age and gender, height and weight, years of education, as well as MS-related information such as EDSS, type of MS, use of assistive device for walking in daily life, and year of diagnosis, will be collected and provided by the centers or via self-report. The participants will be instructed to keep their normal routine but to avoid extraneous physical activity at least 24 hours before the data collection session.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Perceptive Sensitivity | Day 1
  Ratio between participants' reporting frequency and actual variability in motor performance (e.g., gait and sit-to-stand [STS]), referred to as the 'Detection-rate.' Number of pinches is divided by the Coefficient of Variability (in %, of speed or smoothness parameter) in the studied time-window.
Detection Accuracy | Day 1
  Accuracy of detecting naturally occurring variations in self-paced gait and sit-to-stand (STS) performance. Objective change points (events) in speed/smoothness are identified using peak detection algorithms with a predefined threshold to extract only perceptually meaningful speed/smoothness fluctuations. Participants indicate perceived changes using a pinch gesture. A response is classified as correct if it occurs within a ±2-second window of a detected event. Responses outside this window or unmatched with any event are incorrect. Perceptive accuracy is modeled as a binary variable (correct/incorrect) and analyzed using mixed-effects logistic regression to account for repeated measures within subjects.
Correspondence Accuracy | Day 2
  Intra-subject correlation between perceived and actual imposed variations in walking speed or seat height, across different difficulty levels.
  Pearson correlations will study the linear relationship between the exercise difficulty and the reported difficulty. A Fisher Z transformation is carried out on all correlations before further analysis (group level comparisons across participants).
  -Detailed Picture of Each Phase: Average exercise difficulty and reported difficulty are calculated for every 30 s (or 3 STS repetitions). Multiple mixed model analyses are performed on the phases separately, with exercise difficulty and reported difficulty as dependent variables in separate analyses.
  Group (patient versus controls) and time are used as independent variables in all analyses. To control for potential baseline differences in any of the outcome variables exercise and reported difficulty in the last 30 s of the baseline phase are added as covariates in the analyses.

SECONDARY OUTCOMES:
Confidence Rating | Day 1 and 2
  A short structured interview follows the experimental tasks of Day 1 and Day 2, including the following question: "On a scale from 0 to 100, how certain are you that you have been precise/accurate in detecting ongoing variations in your performance? Please mark your confidence level on the presented visual scale". Higher values representing higher confidence (subjective beliefs on their perceptive accuracy).
Perceptive Awareness | Day 1 and 2
  Degree of correspondence between participants' subjective confidence ratings and actual perceptual accuracy in detecting motor performance changes.
  To obtain a crude measure of perceptive awareness, we use two complementary approaches. First, we calculate a confidence-accuracy gap for each participant by subtracting their objective task accuracy from their retrospective confidence rating (in %). Positive values indicate overconfidence, while negative values indicate underconfidence. Second, to assess metacognitive awareness at the group level, we computed the correlation between participants' confidence ratings and their task accuracy. This group-level analysis provides an estimate of whether individuals who were more accurate also tended to be more confident or if there are specific trends differing between groups.
Interoceptive Sensibility | Day 1
  Participants' self-reported (subjective) beliefs about their interoceptive abilities is assessed using the Multidimensional Assessment of Interoceptive Awareness (MAIA-2). This scale is a self-report questionnaire to measure multiple dimensions of interoception: 8 different subscales, each averaging the items scores ranging from 0-5 (higher scores representing higher reported interoceptive abilities).
Proprioceptive Sensibility | Day 1
  Self-reported awareness of body posture consisting of 12 items, and with a total score ranging from 12 to 84, with higher scores representing higher reported postural awareness.
Interoceptive Sensitivity and Attention Questionnaire (ISAQ) | Day 1
  This scale is a self-report measure assessing sensitivity and attention to interoceptive signals. It is divided in 3 subscales: -Sensitivity to neutral bodily sensations (items 1, 3, 5, 8, 9, 11, 13, 15, 17) -Attention to unpleasant bodily sensations (items 6, 10, 14, 16) -Difficulty disengaging from unpleasant bodily sensations (items 2, 4, 7, 12 all reverse scored before summing). Total score ranges from 17-85 but for this study only the first 2 subscales will be considered: 'Sensitivity to neutral bodily sensations' (score range 9-45) and 'Attention to unpleasant bodily sensations' (score range 4-20) with higher scores representing higher reported sensitivity or attention.
6 minutes walking test | Day 1
  The total distance and the distance walked, in meters, minute-by-minute will be recorded during the 6-minutes walking test.

OTHER OUTCOMES:
Visual Analogic Scale for Fatigue | Day 1 and 2
  Self-reported fatigue levels assessed using a Visual Analog Scale (VAS) ranging from 0 ('not at all fatigued') to 10 ('extrimely fatigued'), measured before and after each experimental session (eg. 6MWT or STS experiments).
Hospital Anxiety and Depression Scale (HADS) | Day 1
  A two dimension scale (7 items subscale Depression, 7 items subscale Anxiety) developed to identify depression and anxiety among physically ill patients. Total score: 0-42. Higher scores represent higher Anxiety or depression.
Positive and Negative Affect Schedule (PANAS) | Day 1
  Brief scale to administer to assess positive and negative affect with 2 subscales of 10 items each. Range score is 10-50 for each subscale. Higher scores in each subscale represent higher positive (or negative) affect.
Fatigue Scale for Motor and Cognitive Functions (FSMC) | Day 1
  A 20-item questionnaire assessing how fatigue impact on quality of life. Fatigue severity scores range from 1 (Does not apply at all) to 5 (Applies completely), with higher scores indicating more severe fatigue and greater impact on daily activities.
Dual-Joint Position Test (DJPT) | Day 1
  The Dual-Joint Position Test (clinical test for proprioception) is applied using the second and fourth toes. Both digits move together upward and then downward. Next, they are placed in opposite directions-one up and the other down, and vice versa. Subjects are asked to identify each position with eyes closed. Failure to recognize the toe positions within 10 seconds or more is considered an abnormal response.
Brief Visuospatial Memory Test (BVMDT) | Day 1
  The BVMT-R is a visuospatial memory test, such that participants view a stimulus page for 10 seconds and are asked to draw as many of the figures as possible in their correct location on a separate sheet of paper (6 figures in 6 assigned positions). The participant has 3 attempts, viewing the same figures 3 times. Each attempt can have a maximum score of 12 and the scores are summed together in a total score (0-36).
Symbol Digit Modalities Test (SDMT) | Day 1
  The SDMT is a timed thinking task that involves associating numbers with symbols. Participants will be asked to provide (saying out loud) as many correct numbers as they can within 90 seconds. Score is obtained counting the correct given answers and higher scores represent better cognitive executive functions (ie. information processing speed).
Distance walked index (DWI) | Day 1
  The distance walked index (DWI) will be applied to the distance walked in each minute of the 6-minute walking test performed by the subjects, using the following formula: DWI(%) = ((distance walked at minute n- distance walked at minute 1)/ distance walked at minute 1)*100
Walking speed | Day 1 and 2
  Distance covered per time unit is collected via motion analysis wearable/portable sensors: the anteroposterior distance, divided by the gait cycle duration (two subsequent heel strikes of the same leg), expressed in meter per second.
Walking smoothness | Day 1 and 2
  Harmonic Ratio (HR) is a quantitative measure of gait smoothness, derived from frequency analysis of trunk accelerations, in the antero-posterior direction, during walking.
  It reflects the degree of symmetry and consistency in step-to-step movements: higher HR values indicate a smoother, more coordinated gait, while lower values suggest irregularity or lower smoothness.
Sit-to-Stand speed | Day 1 and 2
  Sit-to-Stand duration is registered via motion analysis wearable/portable sensors: the time to cover the vertical distance represented by the standing-sitting position and expressed in seconds.
Sit-to-Stand Smoothness | Day 1 and 2
  SPARC (SPectral Arclenght) measurement is a measure of the "complexity", or "length", of a movement's frequency spectrum. In particular, it measures the lenght of the curve of the normalized spectrum of the signal (accelleration in the vertical direction) in the frenquency domain. Values of SPARC are of negative value with higher values (closer to 0) representing higher smoothness and lower (more negative) values representing lower smoothness.
COP measures of standing balance | Day 1
  The Test for the Sensory Interaction of Balance will be used to define the proprioceptive interaction on balance: force plates will measure center of pressure (COP) displacement (Area of COP displacement expressed in cm²) in response to standing on a stable and unstable support surface (standard foam pad), with eyes open and closed.
  The degree of increase in COP displacement when applying the foam represents the proprioception quotient (i.e. reliance of body balance on the proprioceptive system). The degree of increase in COP displacement when closing the eyes represents the vision quotient (i.e. reliance of body balance on the visual system).
Rate of Perceived Stability | Day 1
  After each of the four conditions of the Test for the Sensory Interaction of Balance the participant will be asked for a Rate of Perceived Stability, a 1-10 ('completely stable' - 'about to fall') visual analogical scale to rate the perceived balance challenge.
Checklist for Symptoms in Daily life (CSD) | Day 1
  This checklist consists of 39 symptoms that patients can experience in daily life. It measures how often the patients experience the symptoms on a 5-point scale (never, seldom, sometimes, often, very often). Total score ranges from 0 to 156 with higher scores representing higher severity of symptoms in daily life.
Pittsburgh Sleep Quality Index (PSQI) | Day 1
  This scale assesses sleep quality to identify 'good' or 'poor' sleepers, detects the presence of significant sleep disturbance of various types over the past 30 days, and provides an index that can be interpreted by patients, clinicians and researchers. Total score ranges from 0-21 with higher scores identifying higer sleep disturbances.
Brief Pain Inventory (BPI) | Day 1
  The Brief Pain Inventory (BPI) is a self-reported outcome measure that collects the participants' severity of pain and its impact on daily functioning. In particular we consider the 'Severity' subscale which has a total score that can range from 0-10 with higher scores representing higher pain severity.
Modified Fatigue Impact Scale (MFIS) | Day 1
  A 21-item questionnaire assessing the impact of fatigue on physical, cognitive, and psychosocial functioning. Scores can be obtained separately or in total (physical: 0-36; cognitive: 0-40; psychosocial: 0-8; total: 0-80). Higher scores reflect a greater impact of fatigue.
Multiple Sclerosis Walking Scales (MSWS-12) | Day 1
  A 12-item self-reported questionnaire measuring the impact of MS on walking. Scores range from 12 to 60, with higher scores indicating greater walking impairment
Godin Leisure-Time Exercise questionnaire (GLTEQ) | Day 1
  This scale is a self report measure of physical activity. It measures the frequency and intensity of exercise during free time in a typical week. It consists of 3 items and has no upper limit: higher scores represent higher levels of physical activity patricipation.
General Self-Efficacy scale (GSE) | Day 1
  This questionnaire measures self-perception of self-efficacy. The test asks the patients to rate their perceived self-efficacy: to predict their coping abilities. Total score ranges from 10 to 40, with higher scores representing higher self-efficacy.
Control subscale of the Multiple Sclerosis Self-Efficacy scale (MSSE-c) | Day 1
  Subscale of the Multiple Sclerosis Self-Efficacy scale, measuring confidence with managing symptoms and coping with the demands of illness, with a total score ranging from 90 to 900: it consists of 9-item, each item is scored on a Likert-like scale form 10 (very uncertain) to 100 (very certain).
Falls Efficacy Scale International (FES-I) | Day 1
  Subjective report on the concern about falling. It is a 16 items questionnaire with a total score ranging from 16 to 64 (higher scores representing higher concern about falling during activities of daily life)
Timed 25-Foot Walk test (T25-FW) | Day 1
  It is a walking capacity test where the person has to walk as fast as possible, without running, for 7.62 meters. The time needed to complete is recorded in two valid trials. This test will be executed with a flying start (allowing gait accelleration prior to start the timed test).
Expanded Disability Status Scale (EDSS) | Day 1
  It is a classification rate of disability for people with multiple sclerosis ranging from 0 (no disability) to 10 (bedridden due to MS).
Walking Foot Strike Angle | Day 1 and 2
  The dorsiflexion of the feet in the heel strike.
Walking Cadence | Day 1 and 2
  Number of steps made per minute (both legs).
Sit-to-Stand Lean Angle | Day 1 and 2
  The forward trunk inclination a person makes when rising from a seated position to standing: the angle between the vertical axis and the trunk at the point of maximum forward flexion during the sit-to-stand task.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - REVAL, Diepenbeek, Belgium
  - Noorderhart Revalidatie & MS, Overpelt, Belgium
  - Nationaal MS-Centrum Melsbroek, Steenokkerzeel, Belgium

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT07175792/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT07175792/ICF_001.pdf